CLINICAL TRIAL: NCT00178165
Title: Coordinating Center for Enhancing Alzheimer Disease and Related Disorder Caregiving
Brief Title: Coordinating Center for Enhancing ADRD Caregiving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Nursing Research (NINR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG13305-01; NR13269; AG13313; AG13297; AG13289; AG13265; AG13255; AG13305
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Family Caregivers; Dementia; Alzheimer Disease; Randomized Controlled Trial; Intervention Studies
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Drug Delivery Systems

INTERVENTIONS:
Procedure: Skill Training Condition - problem solving training
Procedure: REACH for TLC (Telephone Linked Computer) system

SUMMARY:
Established in 1995, Resources for Enhancing Alzheimer's Caregiver Health (REACH) is a unique, multi-site research program sponsored by the National Institute on Aging (NIA) and the National Institute on Nursing Research (NINR). The primary purpose of REACH is to carry out social and behavioral research on interventions designed to enhance family caregiving for Alzheimer's disease and related disorders. Specifically, REACH has two goals: to test the effectiveness of multiple different interventions and to evaluate the pooled effect of REACH interventions overall. REACH grew out of a National Institute of Health (NIH) initiative that acknowledged the well-documented burdens associated with family caregiving as well as the existence of promising family caregiver interventions reported in the literature.

DETAILED DESCRIPTION:
Six sites (Boston, Birmingham, Memphis, Miami, Palo Alto, and Philadelphia) developed and evaluated a variety of multi-component interventions for family caregivers of persons with Alzheimer's Disease (AD) at the mild or moderate level of impairment. The multi-component interventions implemented across the six sites included: 1) Individual Information and Support strategies, 2) Group Support and Family Systems therapy, 3) Psychoeducational and Skill-based Training approaches, 4) Home-based Environmental interventions,, and 5) Enhanced Technology Support Systems. Although the interventions were derived from diverse theoretical models, they are all consistent with basic health-stress models in which the goal is to change the nature of specific stressors (e.g. problem behavior of the care recipient), their appraisal, and/or the caregivers response to the stressors. All of the REACH interventions were guided by detailed treatment manuals and certification procedures that assured that the interventions were delivered consistently over time at each site. Careful attention was also paid to the issue of treatment integrity. Different strategies were used at each site to induce and assess all three fundamental aspects of treatment integrity: delivery, receipt, and enactment (Burgio, et al., 2001). In addition, because the caregiving experience in race and ethnic minority families is particularly neglected in the field, there was a strong emphasis placed on the inclusion of African American and Hispanic caregivers. Thus, assessments as well as interventions were tailored at each site to meet the needs of culturally diverse racial/ethnic majority and minority populations.

All of the REACH sites shared several common goals, including: 1) designing theory-driven caregiving interventions to test hypotheses about intervention processes and their effect on family caregivers, 2) specifying intervention components that help us understand the pathways through which interventions produce desired outcomes, 3) developing a standardized outcome protocol to assess the impact of different strategies on caregivers and their care recipients within each site and across sites, and 4) creating a common database that would facilitate pooling data across sites. In addition, standard selection criteria were adopted by REACH.

Although REACH has some of the features of a traditional multi-site randomized controlled clinical trial (e.g., random assignment of participants to treatment and control conditions, common database and outcome measures, and identical measurement intervals across sites), it differs on one key dimension-the interventions varied across sites. REACH was designed to examine the feasibility and outcomes of multiple different intervention approaches, rather than to provide definitive information on the efficacy of one specific intervention strategy for enhancing caregiver outcomes. The strength of this approach is that it efficiently yields information about the effectiveness of different approaches to AD caregiving as well as the combined effects of active treatment versus controls, as reported in the planned meta-analysis.

REACH successfully randomized 1222 caregiver/care recipient dyads representing both majority and minority populations to 15 different conditions.

ELIGIBILITY:
CORE CARE RECIPIENT INCLUSION/EXCLUSION CRITERIA

Inclusion criteria:

1. NINCDS -ADRDA Criteria for Alzheimer's Disease and/or DSM IV Criteria for Alzheimer's Disease or other dementia or MMSE score < 23.
2. Functional impairment: presence of two IADL or one ADL impairments.

Exclusion criteria:

1. Any terminal illness with life expectancy < 6 months
2. Active treatment (chemotherapy, radiation therapy) for cancer
3. More than three acute medical hospitalizations in past year (not for psychiatric or Alzheimer's Disease related admission)
4. Schizophrenia (onset of delusions before age 45)
5. Dementia secondary to head trauma (probable)
6. Blindness or deafness if either disability prohibits them from completion of data collection or participation in the interventions
7. MMSE = 0 and bedbound (confined to a bed or chair for > 22 hours per day, for at least 4 of the past 7 days)
8. Planned nursing home admission in 6 months

CORE CAREGIVER INCLUSION/EXCLUSION CRITERIA

Inclusion criteria:

1. Age: 21 years and older
2. Language: site specific, must be competent either orally or written
3. Lives with care recipient
4. Family member
5. Gender: Palo Alto/Los Angeles will only enroll women. All other sites will enroll men and women
6. Must have a telephone
7. At enrollment, plan to remain in area for the duration of the intervention and follow-up
8. Caregiver role of at least 6 months
9. Provides > 4 hours of supervision or direct assistance per day for the care recipient

Exclusion criteria:

1. Any terminal illness with life expectancy < 6 months
2. Active treatment (chemotherapy, radiation therapy) for cancer
3. More than three acute medical hospitalizations in past year
4. Involved in another clinical trial of interventions for caregivers (non drug study)

Second Level Review If the caregiver has been inconsistent with answers or repeated answers, then the interviewer will administer the SPMSQ. The interviewer will then discuss with the PI and coordinate another phone call with the caregiver.

If in the course of the telephone screen the research assistant believes that there may be difficulties for the caregiver regarding travel arrangements, hesitancy to answer questions, or other specific items (site-specific indications), the research assistant will refer to the PI for review.

All potential caregivers will receive a follow-up phone call for second level exclusion from the trial when appropriate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 1996-09; Study Completion 2001-11

PRIMARY OUTCOMES:
The outcomes were assessed 6 months after randomization and included a measure of burden and a measure of depression. Caregiver burden was assessed using the Revised Memory and Behavior Problem Checklist (RMBPC).
Emotional distress was determined by the Center for Epidemiological Studies Depression Scale (CES-D) a global measure of depression.

SECONDARY OUTCOMES:
Long-term care placement of dementia patients and caregiver health and well-being
Use of cognitive enhancement medication
Clinical significance of caregiver interventions in diverse populations

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schulz, Ph.D., Principal Investigator — Professor of Psychiatry and Director, University Center for Social and Urban Research, University of Pittsburgh
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University and Veterans Affairs, Menlo Park, California
  - University of Miami at Miami, Center on Adult Development and Aging, Miami, Florida
  - Thomas Jefferson University at Philadelphia, Center for Applied Research on Aging and Health, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee

REFERENCES:
- [Result] Belle SH, Czaja SJ, Schulz R, Zhang S, Burgio LD, Gitlin LN, Jones R, Mendelsohn AB, Ory MG; REACH Investigators. Using a new taxonomy to combine the uncombinable: integrating results across diverse interventions. Psychol Aging. 2003 Sep;18(3):396-405. doi: 10.1037/0882-7974.18.3.396. PMID 14518803
- [Result] Czaja SJ, Schulz R, Lee CC, Belle SH; REACH Investigators. A methodology for describing and decomposing complex psychosocial and behavioral interventions. Psychol Aging. 2003 Sep;18(3):385-95. doi: 10.1037/0882-7974.18.3.385. PMID 14518802
- [Result] Wisniewski SR, Belle SH, Coon DW, Marcus SM, Ory MG, Burgio LD, Burns R, Schulz R; REACH Investigators. The Resources for Enhancing Alzheimer's Caregiver Health (REACH): project design and baseline characteristics. Psychol Aging. 2003 Sep;18(3):375-84. doi: 10.1037/0882-7974.18.3.375. PMID 14518801
- [Result] Gitlin LN, Belle SH, Burgio LD, Czaja SJ, Mahoney D, Gallagher-Thompson D, Burns R, Hauck WW, Zhang S, Schulz R, Ory MG; REACH Investigators. Effect of multicomponent interventions on caregiver burden and depression: the REACH multisite initiative at 6-month follow-up. Psychol Aging. 2003 Sep;18(3):361-74. doi: 10.1037/0882-7974.18.3.361. PMID 14518800
- [Result] Schulz R, Belle SH, Czaja SJ, Gitlin LN, Wisniewski SR, Ory MG; REACH Investigators. Introduction to the special section on Resources for Enhancing Alzheimer's Caregiver Health (REACH). Psychol Aging. 2003 Sep;18(3):357-60. doi: 10.1037/0882-7974.18.3.357. PMID 14518799
- [Result] Gallagher-Thompson D, Coon DW, Solano N, Ambler C, Rabinowitz Y, Thompson LW. Change in indices of distress among Latino and Anglo female caregivers of elderly relatives with dementia: site-specific results from the REACH national collaborative study. Gerontologist. 2003 Aug;43(4):580-91. doi: 10.1093/geront/43.4.580. PMID 12937336
- [Result] Burgio L, Stevens A, Guy D, Roth DL, Haley WE. Impact of two psychosocial interventions on white and African American family caregivers of individuals with dementia. Gerontologist. 2003 Aug;43(4):568-79. doi: 10.1093/geront/43.4.568. PMID 12937335
- [Result] Mahoney DF, Tarlow BJ, Jones RN. Effects of an automated telephone support system on caregiver burden and anxiety: findings from the REACH for TLC intervention study. Gerontologist. 2003 Aug;43(4):556-67. doi: 10.1093/geront/43.4.556. PMID 12937334
- [Result] Burns R, Nichols LO, Martindale-Adams J, Graney MJ, Lummus A. Primary care interventions for dementia caregivers: 2-year outcomes from the REACH study. Gerontologist. 2003 Aug;43(4):547-55. doi: 10.1093/geront/43.4.547. PMID 12937333
- [Result] Gitlin LN, Winter L, Corcoran M, Dennis MP, Schinfeld S, Hauck WW. Effects of the home environmental skill-building program on the caregiver-care recipient dyad: 6-month outcomes from the Philadelphia REACH Initiative. Gerontologist. 2003 Aug;43(4):532-46. doi: 10.1093/geront/43.4.532. PMID 12937332
- [Result] Eisdorfer C, Czaja SJ, Loewenstein DA, Rubert MP, Arguelles S, Mitrani VB, Szapocznik J. The effect of a family therapy and technology-based intervention on caregiver depression. Gerontologist. 2003 Aug;43(4):521-31. doi: 10.1093/geront/43.4.521. PMID 12937331
- [Result] Schulz R, Burgio L, Burns R, Eisdorfer C, Gallagher-Thompson D, Gitlin LN, Mahoney DF. Resources for Enhancing Alzheimer's Caregiver Health (REACH): overview, site-specific outcomes, and future directions. Gerontologist. 2003 Aug;43(4):514-20. doi: 10.1093/geront/43.4.514. No abstract available. PMID 12937330
- See also: REACH I website- click here for more information about this study — http://www.edc.gsph.pitt.edu/REACH/